CLINICAL TRIAL: NCT01140724
Title: Predicting Perioperative Opioid Adverse Effects and Personalizing Analgesia in Children
Brief Title: Personalizing Perioperative Analgesia in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Senthil Sadhasivam (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY21070173; R01HD089458 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain
Keywords: pain; genes; morphine; respiratory depression; tonsillectomy; children; Opioid adverse effects; Pharmacogenetics of morphine; Pharmacokinetics of morphine; Personalizing analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood is obtained and analyzed for genetic varaiations
Oversight: Data Monitoring Committee: No

SUMMARY:
In the United States alone, each year approximately 5 million children undergo painful surgery, many of them experience serious side-effects with opioids and inadequate pain relief. Safe and effective analgesia is an important unmet critical medical need in children and its continued existence is an important perioperative safety and economic problem. Inadequate pain relief and serious side effects from perioperative opioids occur frequently in up to 50% of children. Morphine, the most commonly used perioperative opioid, has a narrow therapeutic index and large inter-patient variations in analgesic response and serious side effects. Frequent inter-individual variations in responses to morphine have significant clinical and economic impact with inadequate pain relief at one end of the spectrum of responses and serious adverse effects such as respiratory depression at the other end. Much of the inter-individual variability in response to a dose of morphine following surgical procedures can be explained by single nucleotide polymorphisms (SNPs) in a subset of the genes that encode proteins involved in pain mechanisms and opioid pathway.

DETAILED DESCRIPTION:
Measures and Procedures: Participants will receive standard care, standard anesthetic and an intraoperative dose of morphine per the clinical team.

Research procedures will include:

1. Blood draws for genotyping candidate genes and exploratory genes
2. Standardized PACU (post anesthesia care unit) Protocol: Subjective pain assessments: Numerical Rating Scale (NRS) 0 to 10. Objective assessment with FLACC (facial expression; leg movement; activity; cry; and consolability) scale, 0-10.
3. Significant postoperative pain will be managed in the PACU with rescue doses of morphine and opioids by the clinical team. Analgesic interventions and morphine requirements are collected
4. Effects of opioids on pupil measures
5. Respiratory response to 5% carbon dioxide preoperatively and postoperatively (first 350 patients only). Another measure of end tidal carbon dioxide will be implemented when the device is clinically available.
6. Serial blood draws for morphine pharmacokinetic modeling (through subject #351).
7. Opioid adverse effects in PACU and at home.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls,
* 3-15 years of age,
* all races,
* American Society of Anesthesiologists (ASA) physical status 1,2, and 3,
* children with history of significant snoring suggestive of obstructive sleep apnea (OSA),
* Scheduled for tonsillectomy (T) or tonsillectomy and adenoidectomy (T and A).

Exclusion Criteria:

* allergic to study medications
* developmental delay,
* liver and renal diseases,
* preoperative pain requiring analgesics,
* children who have problems with pupil or pupillary reaction due to disease
* preoperative medications influencing pupillary size
* non-English speaking participants and families
* Body Mass Index ≥30
* Participants undergoing additional procedures during surgery
* Children with certain cardiac conditions
* Children with severe lung disease
* Children with a history of seizures currently treated on medication
* Children with psychiatric/psychological conditions for which patient currently takes medication

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, 3-15 years of age, undergoing tonsillectomy or adenotonsillectomy at the Riley Hospital for Children, who have consented to participate in an observational clinical study as approved by the IU IRB, protocol # 1707325115.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Look at polymorphisms in genes that regulate pain perception, opioid transport and opioid receptor signaling to see if there is a higher susceptibility to pain and morphine requirement. | After tonsillectomy surgery (duration of post anesthesia care unit stay)
  Look at polymorphisms in genes that regulate pain perception, opioid transport and opioid receptor signaling to see if there is a relationship to more pain and need for a higher morphine requirement.

SECONDARY OUTCOMES:
Evaluate relationship of pupil reaction and response to 5% carbon dioxide to adverse effects of morphine | After tonsillectomy surgery (duration of post anesthesia care unit stay)

OTHER OUTCOMES:
Evaluate contribution of polymorphisms in genes to variability in codeine response in children with CYP2D6 genotypes predictive of extensive metabolizer or ultra-extensive metabolizer phenotypes | During tonsilectomies
  Evaluate contribution of polymorphisms in genes that regulate pain perception, opioid transport and opioid receptor signaling to variability in codeine response in children with CYP2D6 genotypes predictive of extensive metabolizer or ultra-extensive metabolizer phenotypes
Evaluate whether machine learning techniques can be used to predict pain response, opioid responses and morphine usage requirements in patients | After tonsilectomy surgery data collection
  Evaluate whether machine learning techniques can be used to predict pain response, opioid responses and morphine usage requirements in patients solely using information extracted from the medical record as well as in combination with other genetic information

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, MPH, Principal Investigator — University of Pittsburgh, UPMC
Locations (1):
- UPMC Children's Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Packiasabapathy S, Zhang X, Ding L, Aruldhas BW, Pawale D, Sadhasivam S. Quantitative Pupillometry as a Predictor of Pediatric Postoperative Opioid-Induced Respiratory Depression. Anesth Analg. 2021 Oct 1;133(4):991-999. doi: 10.1213/ANE.0000000000005579. PMID 34029273
- [Derived] Hahn D, Fukuda T, Euteneuer JC, Mizuno T, Vinks AA, Sadhasivam S, Emoto C. Influence of MRP3 Genetics and Hepatic Expression Ontogeny for Morphine Disposition in Neonatal and Pediatric Patients. J Clin Pharmacol. 2020 Aug;60(8):992-998. doi: 10.1002/jcph.1592. Epub 2020 Feb 24. PMID 32090339
- [Derived] Chidambaran V, Venkatasubramanian R, Zhang X, Martin LJ, Niu J, Mizuno T, Fukuda T, Meller J, Vinks AA, Sadhasivam S. ABCC3 genetic variants are associated with postoperative morphine-induced respiratory depression and morphine pharmacokinetics in children. Pharmacogenomics J. 2017 Mar;17(2):162-169. doi: 10.1038/tpj.2015.98. Epub 2016 Jan 26. PMID 26810133
- [Derived] Sadhasivam S, Zhang X, Chidambaran V, Mavi J, Pilipenko V, Mersha TB, Meller J, Kaufman KM, Martin LJ, McAuliffe J. Novel associations between FAAH genetic variants and postoperative central opioid-related adverse effects. Pharmacogenomics J. 2015 Oct;15(5):436-42. doi: 10.1038/tpj.2014.79. Epub 2015 Jan 6. PMID 25558980
- [Derived] Sadhasivam S, Chidambaran V, Olbrecht VA, Costandi A, Clay S, Prows CA, Zhang X, Martin LJ. Opioid-related adverse effects in children undergoing surgery: unequal burden on younger girls with higher doses of opioids. Pain Med. 2015 May;16(5):985-97. doi: 10.1111/pme.12660. Epub 2014 Dec 17. PMID 25521773
- [Derived] Sadhasivam S, Chidambaran V, Olbrecht VA, Esslinger HR, Zhang K, Zhang X, Martin LJ. Genetics of pain perception, COMT and postoperative pain management in children. Pharmacogenomics. 2014 Feb;15(3):277-84. doi: 10.2217/pgs.13.248. PMID 24533707
- [Derived] Prows CA, Zhang X, Huth MM, Zhang K, Saldana SN, Daraiseh NM, Esslinger HR, Freeman E, Greinwald JH, Martin LJ, Sadhasivam S. Codeine-related adverse drug reactions in children following tonsillectomy: a prospective study. Laryngoscope. 2014 May;124(5):1242-50. doi: 10.1002/lary.24455. Epub 2013 Nov 13. PMID 24122716
- [Derived] Sadhasivam S, Krekels EH, Chidambaran V, Esslinger HR, Ngamprasertwong P, Zhang K, Fukuda T, Vinks AA. Morphine clearance in children: does race or genetics matter? J Opioid Manag. 2012 Jul-Aug;8(4):217-26. doi: 10.5055/jom.2012.0119. PMID 22941849
- [Derived] Sadhasivam S, Chidambaran V, Ngamprasertwong P, Esslinger HR, Prows C, Zhang X, Martin LJ, McAuliffe J. Race and unequal burden of perioperative pain and opioid related adverse effects in children. Pediatrics. 2012 May;129(5):832-8. doi: 10.1542/peds.2011-2607. Epub 2012 Apr 23. PMID 22529273